CLINICAL TRIAL: NCT04139889
Title: The Diagnosis of Laryngeal Lesions Using the Probe-based Confocal Laser Endomicroscopy in Vivo
Brief Title: Diagnosis of Laryngeal Lesions Using the Probe-based Confocal Laser Endomicroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 20170601
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Laryngeal Leiomyoma; Probe-based Confocal Laser Endomicroscopy
Keywords: Probe-based confocal laser endomicroscopy; Optical biopsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- normal mucosa: Flat and relatively uniform polygonal epithelial cells with alternating dark and light bands were noted in pCLE images of normal mucosa after intravenous injecting 10% fluorescein.
  Interventions: Diagnostic Test: Confocal Laser Endomicroscopy
- non-malignant lesions: An unorganized tissue architecture, irregular cells (difference of cell shape, color and size), slightly intensified fluorescein leakage, and vessels not assessable were found in the lymphoid hyperplasia of non-malignant lesions after intravenous injecting 10% fluorescein.
  Interventions: Diagnostic Test: Confocal Laser Endomicroscopy
- malignant lesions: pCLE images of malignant lesions were associated with crowded unorganized tissue architecture (a dark-gray background without identification of mucosal structures), irregular cells like cell clusters, amplified fluorescein leakage, and irregular vessels changes after intravenous injecting 10% fluorescein.
  Interventions: Diagnostic Test: Confocal Laser Endomicroscopy

INTERVENTIONS:
Diagnostic Test: Confocal Laser Endomicroscopy — Confocal laser microendoscopy (CLE) as a new non-invasive imaging technique can be used for "optical biopsy", which can perform real-time microscopic information of tissue in vivo at cellular level with resolutions up to 1μm and magnifications up to 1000 times. CLE is now being increasingly used with very promising results in gastroenterology, especially in the diagnostic investigation of Barret's esophagus, stomach cancer, colorectal cancer and various lesions of the biliary tract. With an intravenous injection of fluorescein, probe-based CLE (pCLE: GastroFlex probe with the Cellvizio laser system, Mauna Technologies, Paris, France) allows us to view the interstitial spaces, cells, and small capillaries in a window of 240 μm and to a depth of 60 μm.

SUMMARY:
To evaluate the diagnosis of laryngeal lesions using the Probe-based Confocal Laser Endomicroscopy in vivo.

DETAILED DESCRIPTION:
In this study, we will conduct in-vivo confocal laser endoscopic imaging studies of laryngeal and precancerous lesions to explore the value of pCLE in the diagnosis of laryngeal cancers.

ELIGIBILITY:
Inclusion Criteria:

1. 18≤Male or female age ≤85 years old;
2. patients with vocal cord lesions founded by white light laryngoscope and needed to perform laryngeal microsurgery;
3. Willing and able to comply with study procedures and provide written informed consent to participate in the study.

Exclusion Criteria:

1. Male or female <18 years old, or Male or female >85 years;
2. The patient has abnormal blood or coagulation function, and there is a risk of bleeding during the examination;
3. The patient has severe cardiopulmonary function or liver and kidney dysfunction and cannot tolerate surgery.
4. The patient has a history of allergies to drugs or food.
5. The patient has a positive serotonin sodium allergy test and is allergic to sodium fluorescein;
6. Lactation or pregnant women.
7. Refusal to sign the informed consent form.
8. Others who do not take this test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with suspicious unidentified lesions were collected in this study in Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, who need to be underwent microscopic laryngoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-21 (Estimated)

PRIMARY OUTCOMES:
pCLE diagnostic classification | 6 months
  Evaluation of pCLE diagnostic performance for the diagnosis of Laryngeal Lesions when associated with other diagnostic information.

SECONDARY OUTCOMES:
the image analysis by machine learning | 6 months
  Quantitative image features are calculated in the pCLE images by machine learning

CONTACTS AND LOCATIONS:
Overall Officials: Huawei Li, PhD &MD, Study Chair — Otorhinolaryngology Department of Eye & ENT Hospital, Fudan University
Locations (1):
- Otorhinolaryngology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No